CLINICAL TRIAL: NCT02123134
Title: A Multicenter, Double-blind, Placebo-controlled Safety Study of ATX-101 (Deoxycholic Acid) Injection for the Reduction of Localized Subcutaneous Fat in the Submental Area in Subjects 65 to 75 Years of Age
Brief Title: Safety Study of Deoxycholic Acid for the Reduction of Localized Subcutaneous Fat in the Submental Area in Subjects 65 to 75 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kythera Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATX-101-13-28
Record Dates: First submitted 2014-04-22; First posted 2014-04-25 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-01

CONDITIONS: Moderate to Severe Convexity of Submental Fat; Safety; Efficacy
MeSH Terms: interventions — Deoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo administered in 0.2 mL subcutaneous (SC) injections, up to 10 milliliters (mL) per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments.
  Interventions: Drug: Placebo
- ATX-101 deoxycholic acid injection (Experimental): Participants received deoxycholic acid 2 mg/cm^2 administered in 0.2 mL SC injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments.
  Interventions: Drug: ATX-101

INTERVENTIONS:
Drug: ATX-101 — Formulated as an injectable solution containing deoxycholic acid at a concentration of 10 mg/mL.
  Other Names: deoxycholic acid
  Arms: ATX-101 deoxycholic acid injection
Drug: Placebo — Phosphate buffered saline placebo for injection
  Arms: Placebo

SUMMARY:
The objectives of this study are to explore the safety and efficacy of subcutaneous injections of Deoxycholic Acid relative to placebo, in the submental area of participants who are 65 to 75 years old.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 65 to 75 years of age
* Stable Body Weight
* Dissatisfaction with the submental area expressed by participants
* Acceptable volume of submental fat graded by clinician
* BMI of ≤40.0 kg/m^2
* Signed informed consent (ICF)
* SMF rating of 2 or 3 by clinician and patient

Exclusion Criteria:

* No prior intervention for submental fat (SMF) (eg liposuction, surgery or lipolytic agents)
* Absence of clinically significant health problems
* Anatomical features for which reduction in SMF may result in aesthetically unacceptable outcome, judged by clinician
* History of trauma associated with the chin or neck areas that in the judgment of the investigator may affect evaluation of safety or efficacy
* Body mass index of ≥40.0 kg/m^2

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Beddingfield, III, MD, PhD, Study Director — Sponsor GmbH
Locations (6):
- United States (6):
  - Birmingham, Alabama
  - Los Angeles, California
  - Bradenton, Florida
  - Metairie, Louisiana
  - White Plains, New York
  - Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 55 subjects were randomized to either ATX-101 or placebo at a ratio of 1:1. A total of 28 subjects received ATX-101 and 26 subjects received placebo; 1 subject (803-003) was randomized to placebo but was not treated with placebo.
Groups:
- ATX-101 (Deoxycholic Acid) Injection: Participants received deoxycholic acid 2 mg/cm^2 administered in 0.2 mL subcutaneous (SC) injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments.
Period: Overall Study
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Started | 28 | 27
Completed | 25 | 24
Not Completed | 3 | 3
Not completed — Withdrawal of consent | 3 | 2
Not completed — Administrative decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (2.76) | 67.7 (2.30) | 67.9 (2.53)
Age, Customized [Count of Participants; unit: Participants]
  65-69 years | 22 | 22 | 44
  70-75 years | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 27 | 25 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 25 | 25 | 50
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick skin type is a numerical classification schema for different skin types and tanning abilities. TYPE 1: Pale white skin, blue/hazel eyes, blond/red hair, always burns, never tans. TYPE 2: Fair skin, blue eyes, burns easily, tans poorly. TYPE 3: Darker white skin, tans after initial burn. TYPE 4: Light brown skin, burns minimally, tans easily. TYPE 5: Brown skin, rarely burns, tans darkly easily. TYPE 6: Dark brown or black skin, never burns, always tans darkly.
  Participants
    I | 0 | 1 | 1
    II | 15 | 10 | 25
    III | 7 | 12 | 19
    IV | 2 | 1 | 3
    V | 3 | 2 | 5
    VI | 1 | 1 | 2
Weight [Mean (Standard Deviation); unit: kg] | 77.44 (14.170) | 84.10 (14.070) | 80.71 (14.388)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.27 (4.207) | 30.72 (4.694) | 29.98 (4.471)
Body mass index category [Count of Participants; unit: Participants]
  Less than 30 kg/m^2 | 15 | 13 | 28
  30 kg/m^2 or greater | 13 | 14 | 27
Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) score [Count of Participants; unit: Participants] — The investigator evaluated the participant's chin and neck area using the Clinician-Reported Submental Fat Rating Scale (a 5-point scale) where: 0=absent submental convexity (best) to 4= extreme submental convexity (worst).
  Participants
    0 | 0 | 0 | 0
    1 | 0 | 0 | 0
    2 | 5 | 6 | 11
    3 | 23 | 21 | 44
    4 | 0 | 0 | 0
Patient-Reported Submental Fat Rating Scale (PR-SMFRS) score [Count of Participants; unit: Participants] — The participant evaluated their chin and neck area using the Patient-Reported Submental Fat Rating Scale (a 5-point scale) where: 0=no chin fat at all (best) to 4= a very large amount of chin fat (worst).
  Participants
    0 | 0 | 0 | 0
    1 | 0 | 0 | 0
    2 | 23 | 19 | 42
    3 | 5 | 8 | 13
    4 | 0 | 0 | 0
Submental Skin Laxity Grade (SMSLG) [Count of Participants; unit: Participants] — The SMSLG is an integration of three features: skin wrinkling, adherence to underlying neck structures (bone and muscle) and redundancy (horizontal and vertical folds). Each grade (1=none, 2=mild, 3=moderate and 4=severe) defines the maximal allowed limit for skin wrinkling, adherence to underlying structures and redundancy.
  Participants
    None | 0 | 1 | 1
    Mild | 8 | 6 | 14
    Moderate | 20 | 20 | 40
    Severe | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least a 1-Grade Reduction (Improvement) at 12 Weeks From Last Treatment Based on Both the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) and Patient-Reported Submental Fat Rating Scale (PR-SMFRS) Assessments
Description: The investigator evaluated the participant's chin and neck area using the Clinician-Reported Submental Fat Rating Scale (a 5-point scale) where: 0=absent submental convexity (best) to 4= extreme submental convexity (worst).
  The participant evaluated their chin and neck area using the Patient-Reported Submental Fat Rating Scale (a 5-point scale) where: 0=no chin fat at all (best) to 4= a very large amount of chin fat (worst).
Time Frame: Baseline and up to Week 32 (12 weeks after last treatment)
Population: Intent-to treat (ITT) population included all randomized participants, whether or not they received the assigned study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Number analyzed (Participants) | 25 | 24
percentage of participants | 68.0 [49.7 to 86.3] | 25.0 [7.7 to 42.3]

2. Primary Outcome: Percentage of Participants With at Least a 2-Grade Reduction (Improvement) at 12 Weeks From Last Treatment Based on Both the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) and Patient-Reported Submental Fat Rating Scale (PR-SMFRS) Assessments
Description: as for outcome 1
Time Frame: Baseline and up to Week 32 (12 weeks after last treatment)
Population: ITT population included all randomized participants, whether or not they received the assigned study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Number analyzed (Participants) | 25 | 24
percentage of participants | 8.0 [0.0 to 18.6] | 4.2 [0.0 to 12.2]

3. Primary Outcome: Percentage of Participants With at Least a 1-Grade Reduction (Improvement) at 12 Weeks From Last Treatment Based on the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS)
Description: The investigator evaluated the participant's chin and neck area using the CR-SMFRS 5-point scale where: 0=absent submental convexity (best) to 4= extreme submental convexity (worst).
Time Frame: Baseline and up to Week 32 (12 weeks after last treatment)
Population: ITT population included all randomized participants, whether or not they received the assigned study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Number analyzed (Participants) | 25 | 24
percentage of participants | 84.0 [69.6 to 98.4] | 41.7 [21.9 to 61.4]

4. Primary Outcome: Percentage of Participants With at Least a 2-Grade Reduction (Improvement) at 12 Weeks From Last Treatment Based on the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS)
Description: as for outcome 3
Time Frame: Baseline and up to Week 32 (12 weeks after last treatment)
Population: ITT population included all randomized participants, whether or not they received the assigned study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Number analyzed (Participants) | 25 | 24
percentage of participants | 60.0 [40.8 to 79.2] | 12.5 [0.0 to 25.7]

5. Primary Outcome: Percentage of Participants With at Least a 1-Grade Reduction (Improvement) at 12 Weeks From Last Treatment Based on the Patient-Reported Submental Fat Rating Scale (PR-SMFRS)
Description: The participant evaluated their chin and neck area using the PR-SMFRS 5-point scale where: 0=no chin fat at all (best) to 4= a very large amount of chin fat (worst).
Time Frame: Baseline and up to Week 32 (12 weeks after last treatment)
Population: ITT population included all randomized participants, whether or not they received the assigned study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Number analyzed (Participants) | 25 | 24
percentage of participants | 80.0 [64.3 to 95.7] | 45.8 [25.9 to 65.8]

6. Primary Outcome: Percentage of Participants With at Least a 2-Grade Reduction (Improvement) at 12 Weeks From Last Treatment Based on the Patient-Reported Submental Fat Rating Scale (PR-SMFRS)
Description: as for outcome 5
Time Frame: Baseline and up to Week 32 (12 weeks after last treatment)
Population: ITT population included all randomized participants, whether or not they received the assigned study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Number analyzed (Participants) | 25 | 24
percentage of participants | 20.0 [4.3 to 35.7] | 20.8 [4.6 to 37.1]

7. Primary Outcome: Change From Baseline in Submental Skin Laxity Grade Scale (SMSLG)
Description: The SMSLG is an integration of three features: skin wrinkling, adherence to underlying neck structures (bone and muscle) and redundancy (horizontal and vertical folds). Each grade (1=none, 2=mild, 3=moderate and 4=severe) defines the maximal allowed limit for skin wrinkling, adherence to underlying structures and redundancy.
Time Frame: Baseline and up to Week 32 (12 weeks after last treatment)
Population: ITT population included all randomized participants, whether or not they received the assigned study drug.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Number analyzed (Participants) | 25 | 24
scores on a scale | -0.5 (0.65) | -0.1 (0.45)

ADVERSE EVENTS:
Time Frame: Up to 32 Weeks
Description: Safety population included all randomized participants who received at least 1 injection of study drug.
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/26
Other Adverse Events (participants affected / at risk) | 28/28 | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATX-101 (Deoxycholic Acid) Injection (N=28) | Placebo (N=26)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATX-101 (Deoxycholic Acid) Injection (N=28) | Placebo (N=26)
Injection site bruising (General disorders) | 20 (42) | 15 (35)
Injection site pain (General disorders) | 20 (44) | 3 (6)
Injection site swelling (General disorders) | 17 (38) | 15 (54)
Injection site anaesthesia (General disorders) | 14 (16) | 0 (0)
Injection site nodule (General disorders) | 8 (8) | 3 (3)
Injection site oedema (General disorders) | 5 (14) | 0 (0)
Injection site erythema (General disorders) | 4 (9) | 3 (4)
Injection site induration (General disorders) | 4 (7) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Skin tightness (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.